CLINICAL TRIAL: NCT04906434
Title: A Phase 1, Open-Label Study of ABSK-011 to Assess Safety, Tolerability, and Pharmacokinetics in Patients With Advanced Solid Tumors
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of ABSK-011 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABSK-011-101
Record Dates: First submitted 2021-04-21; First posted 2021-05-28 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Liver Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABSK-011 (Experimental): During the escalation part, all patients will first receive a single dose ABSK-011 (run-in period) at Day -2 and be followed by a 1-day off (2 days in all for run-in period) to access the PK of single-dose. Then, patients will continuously receive ABSK-011 once daily (QD) or twice daily (BID) in repeated 28-day cycles. Dose escalation will employ a "3+3" design except for the patient in the accelerated titration cohort. In expansion part, patients will be treated at the selected RDE dose level.
  Interventions: Drug: ABSK-011

INTERVENTIONS:
Drug: ABSK-011 — During the escalation part, the administration of oral ABSK-011 will be guided by "3+3"design based on safety data collected until a maximum tolerated dose (MTD) has been identified. The first dose level will be administered as QD, and different dosing frequencies (e.g., BID) may be explored in subsequent doses depending on emerging safety and pharmacokinetic data. A separate food effect cohort may be conducted. In expansion part, patients will be treated at the selected RDE dose level.

SUMMARY:
This is an open-label phase 1 study with an escalation part and an expansion part.

DETAILED DESCRIPTION:
The escalation part will evaluate the safety, tolerability, PK and recommended dose of expansion (RDE) of oral ABSK-011 in patients with advanced solid tumors. The expansion part of oral ABSK-011 at RDE will be followed for further evaluating safety and tolerability in patients with FGF19 overexpression advanced HCC. Preliminary antitumor activity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 ~ 75 (include both ends, or other age range required by local regulations or IRB).
2. Escalation Part: Patients must have histological or cytological confirmed advanced solid tumors that have progressed on or intolerant to standard therapy or whom no standard therapy exists; and patients with advanced HCC must satisfy:

   1. BCLC stage B or C and Child-Pugh score 5~6
   2. Patient must provide archived tissue sample or biopsy for FGF19 overexpression central lab testing

   Expansion Part: patients must have histological or cytological confirmed, BCLC stage B or C HCC, and have progressed on or intolerant to or have refused to receive or have no access to receive first line systemic therapy (by local guideline/regulation) and is unsuitable for other standard therapy(ies) (by local guideline/regulation) against HCC, and must satisfy:
   1. Patient must provide archived tissue sample or biopsy for FGF19 overexpression central lab testing, and the result must be positive
   2. Patient must have at least 1 measurable lesion (RECIST V1.1)
   3. Child-Pugh score 5~7 without hepatic encephalopathy, no clinically apparent ascites or require medical intervention
3. ECOG performance status 0~1
4. Life expectancy ≥ 3 months
5. Adequate organ function and bone marrow function as indicated by the following screening assessments performed within 14 days prior to the first dose of study drug (without blood transfusion or medication with stimulation factors within 14 days before 1st dose):

   1. Absolute neutrophil count (ANC) ≥1.5×109/L
   2. Platelet count (PLT) ≥75×109/L
   3. Hemoglobin (Hb) ≥80 g/L
   4. Total bilirubin (TBIL) ≤1.5×ULN
   5. Aspartate transaminase (AST) and alanine transaminase (ALT), ≤3×ULN (for patient with liver metastasis in escalation part or patient in expansion part: AST and AST ≤5×ULN)
   6. Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Crcl) ≥50 mL/min based on Cockcroft-Gault formula
6. Patients with HBV infection should follow local clinical practice and anti-HBV therapy should be performed to ensure adequate viral suppression (HBV-DNA < 10000 IU/mL or equivalent copies/mL prior to enrollment). Patients are examined every cycle to monitor HBV-DNA levels. If virus reactivation occurred for patients without anti-viral treatment when enrolled, anti-HBV therapy will be started following local practice.
7. Non-surgically sterilized male or female patients of childbearing potential must agree to use effective methods of birth control during the study and for up to 6 months after the last dose of study drug. Non-surgically sterilized female patients of childbearing potential must in non-lactation period, and have a negative β-HCG test result within 7 days before first administration.
8. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.

Exclusion Criteria:

1. Known allergy or hypersensitivity to any component of the investigational drug product.
2. Previous treatment with FGFR4 or pan-FGFR pathway inhibitors (pan-FGFR inhibitors should be confirmed with the sponsor).
3. Has a known second primary malignancy required active treatment.
4. Has a known active central nervous system (CNS) metastases (if stable disease after treatment, free from or daily dexamethasone <10 mg or other equivalent glucocorticoids can be enrolled).
5. Liver tumor volume accounts for ≥50% of the whole liver.
6. Inability to take oral medication or other factors significant preclude adequate absorption of oral medication, such as previously received total gastrectomy, residual gastric dysfunction after subtotal gastrectomy, short bowel syndrome after small bowel resection, active diarrhea required drug treatment, etc.
7. Severe irritable bowel syndrome requires drug therapy.
8. Prior organ transplantation requires anti-rejection drug therapy.
9. Previous anti-cancer therapy prior to initiation of study treatment: major surgery (except palliative therapy), radiotherapy (bone-marrow exposure >30%), routine chemotherapy <4 weeks (chemotherapy with nitrosourea or mitomycin <6 weeks); oral chemotherapy, endocrine therapy, molecular targeted therapy or immunotherapy within ≤ 5 half-life or ≤ 4 weeks (whichever is shorter).
10. Prior toxicities from chemotherapy, radiotherapy, and other anti-cancer therapies, including immunotherapy that have not regressed to Grade ≤1 severity (CTCAE v5.0) with the exception of which inclusion criteria allowed, alopecia, vitiligo and neurotoxicity Grade ≤2 that investigator believe don't affect safety assessment.
11. Concomitant use of strong inhibitors or inducers of CYP3A4 (include grapefruit juice, grapefruit hybrids, pomegranates, starfruit, pomelos, Seville oranges or juice or products) within at least 14 day prior to the first dose of the study drug.
12. Impaired cardiac function or clinically significant cardiac disease, including any one of the following:

    1. New York Heart Association class III or IV congestive heart failure, unstable angina, or myocardial infarction within 6 months before administration of the study drug;
    2. Clinically significant cardiac arrhythmia requiring active therapy;
    3. Uncontrolled hypertension;
    4. Left ventricle ejection fraction<50%
    5. Prolongation of QTcF (average of three times of examine, male > 450 ms, female > 470 ms) (Note: QTc interval corrected by Frederica's formula) at screening, and other ECG abnormalities with clinical significant by the judge of the investigator.
13. Active infection or unexplained fever > 38.5℃.
14. Active or record of gastrointestinal bleeding within 6 months (e.g. esophageal varices or ulcer bleeding).
15. Patients with active HCV infection (HCV-RNA>103 copies/mL or following local clinical practice) and require concomitant anti-HCV therapy during the study; or HBV HCV co-infection.
16. History of immunodeficiency, including HIV serum test positive, or other acquired/congenital immunodeficiency disease, or active tuberculosis.
17. Any other clinically significant comorbidities, such as respiratory, metabolic, congenital, endocrine or central nervous system disease, or any other medical conditions, mental disturbances or social determinants, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.
18. Combined with portal vein tumor thrombus of type IV.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | From the starting dosing of study drug to the end of Cycle 1 (each cycle is 28 days) in escalation Part
  Incidence of dose-limiting toxicities (DLTs) in Cycle 1
Incidence and severity of AEs, AESIs and SAEs | 30 days after last administration, an average of one half year
  Incidence and severity of adverse events (AEs), adverse events of special interest (AESIs) and serious adverse events (SAEs) (Common Terminology Criteria for Adverse Events, CTCAE 5.0)
dose reduction or discontinuation | through study completion, an average of one half year
  dose reduction or discontinuation of study drug due to toxicity
physical examinations changes from baseline | through study completion, an average of one half year
  BMI
ECOG performance status | through study completion, an average of one half year
  ECOG performance status
electrocardiograms (ECGs) | through study completion, an average of one half year
  QTc
echocardiograms changes from baseline | through study completion, an average of one half year
  EF%
vital signs changes from baseline | through study completion, an average of one half year
  Temperature
vital signs changes from baseline | through study completion, an average of one half year
  pulse
vital signs changes from baseline | through study completion, an average of one half year
  blood pressure

SECONDARY OUTCOMES:
Cmax | the end of Cycle 1 Day15 (each cycle is 28 days)
  maximum observed concentration (Cmax)
Tmax | the end of Cycle 1 Day15 (each cycle is 28 days)
  time to maximum observed concentration (Tmax)
AUC | the end of Cycle 1 Day15 (each cycle is 28 days)
  area under the concentration-time curve (AUC)
t1/2β | the end of Cycle 1 Day15 (each cycle is 28 days)
  elimination half-life (t1/2β)
Vz/F | the end of Cycle 1 Day15 (each cycle is 28 days)
  apparent volume of distribution (Vz/F)
CL/F | the end of Cycle 1 Day15 (each cycle is 28 days)
  apparent oral clearance (CL/F)
Css_max | the end of Cycle 1 Day15 (each cycle is 28 days)
  maximum observed concentration of steady-state (Css_max)
Css_min | the end of Cycle 1 Day15 (each cycle is 28 days)
  minimum observed concentration of steady-state (Css_min)
AUCss | the end of Cycle 1 Day15 (each cycle is 28 days)
  area under the concentration-time curve of steady-state (AUCss)
Rac | the end of Cycle 1 Day15 (each cycle is 28 days)
  accumulation rate (Rac)
ORR | throughout study completion, on average of half year
  Evaluate the preliminary antitumor activity in patients with FGF19 overexpression advanced HCC and in patients with other types of advanced solid tumor
DoR | throughout study completion, on average of half year
  Duration of response (DoR): time from [PR] or [CR] to disease progression
DCR | throughout study completion, on average of half year
  Disease control rate (DCR): DCR = [CR] +[PR] + stable disease [SD]
PFS | throughout study completion, on average of half year
  Progression-free survival (PFS): time from the first day receive study drug to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Doctor, Principal Investigator — Tongji Hospital
Locations (32):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- China (24):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The Fifth Medical Center of the General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen Memorial Hospital, Guangzhou, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - Weifang People's Hospital, Weifang, Hebei
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Suzhou University Affiliated Second Hospital, Suzhou, Jiangsu
  - Tonghua Central Hospital, Tonghua, Jilin
  - Shengjing Hospital of China medical university, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Ningbo Huamei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang
- Taiwan (2):
  - National Cheng Kung University Hospitals, Tainan
  - Nation Taiwan University Hospital, Taipei